CLINICAL TRIAL: NCT03981081
Title: Eosinophil-guided Prednisone Administration in COPD Exacerbation Requiring Ventilatory Support
Brief Title: Prednisone Reduction in ICU Patients With COPD Exacerbation
Acronym: EoPred-ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Universitaire Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Fekri Abroug, Professor, ICU Head, Hôpital Universitaire Fattouma Bourguiba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01RM2019
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Copd Exacerbation Acute; Mechanical Ventilation
Keywords: COPD; Acute hypercapnic respiratory failure; Steroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, open-label, parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eosinophil-guided group (Experimental): patients will receive prednisone at a dose of 1mg/kg/day for up to 5 days or during the hospital stay if less than 5 days, only if the eosinophil count is> 2%
  Interventions: Drug: Prednisone
- control group (Active Comparator): a treatment based on prednisone at a daily dose of 1 mg/kg will be routinely administered for a maximum of 5 days, or during the hospital stay, if it is less than 5 days
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Corticosteroid treatment is taken in the morning in patients with NIV, and through the gastric tube in intubated patients

SUMMARY:
The aim of this multicenter, investigator-initiated, prospective, randomized, open-label, non-inferiority study is to evaluate a prednisone prescribing strategy, guided by eosinophil blood count compared to the standard (systematic) administration of corticosteroids, in patients with COPD exacerbation requiring ventilatory support.

Patients fulfilling inclusion criteria and consenting to participate in the study, will be randomized through a random table generated electronically, to eosinophil-guided group or to control group.

In the eosinophil-guided group, prednisone (1mg/kg/day for up to 5 days or during the hospital stay if less than 5 days) is administered only if the eosinophil count is >2%. If blood eosinophil count is ≤2%, no corticosteroids are given. In the control group: a treatment based on prednisone at a daily dose of 1 mg/kg will be routinely administered for a maximum of 5 days, or during the hospital stay, if it is less than 5 days. Corticosteroid treatment is taken in the morning in patients with NIV, and through the gastric tube in intubated patients.

The hypothesis tested is a non-inferiority of the "eosinophil-guided strategy" compared to the standard strategy, with less exposure to corticosteroids.

The primary endpoint is the proportion of unventilated patients at day 6 which is set to 50% in the control group. A pre-specified difference <10% would be a non-inferiority margin.

Secondary endpoints are: Number of ICU days alive without ventilatory support within 28 days after recruitment, length of stay in intensive care Unit, the intubation rate in patients initially under NIV, Mortality in the ICU, Hospital mortality.

Safety: New onset of diabetes or worsening of diabetes requiring the start or the increase in insulin therapy, Upper gastrointestinal bleeding (2 g drop of Hb requiring blood transfusion or fibroscopy), Uncontrolled hypertensive crisis requiring the introduction of new antihypertensives, ICU-acquired neuromyopathy, Nosocomial infection, Relapse rate / recurrence defined respectively by the rate of a new hospital consultation and/or admission in the week or the month following index hospitalization.

Sample size calculation: In a non-inferiority study, with an incidence of the event (no ventilation at D6) of 50% in the control group ( with 10% of acceptable difference for non-inferiority), a power of 80% and alpha error <0.05, it would take 86 patients per arm by anticipating 2% of lost sight.

DETAILED DESCRIPTION:
The aim of this multicenter, investigator-initiated, prospective, randomized, open-label, non-inferiority study is to evaluate a prednisone prescribing strategy guided by eosinophil blood count compared to the standard (systematic) administration of corticosteroids in patients with COPD exacerbation requiring ventilatory support,.

Consecutive patients admitted to the ICU with hypercapnic respiratory failure consecutive to COPD exacerbation, and requiring ventilatory support with non-invasive or invasive mechanical ventilation, will be considered for inclusion in the study.

Patients fulfilling inclusion criteria and consenting to participate in the study, will be randomized through a random table generated electronically, to eosinophil-guided group or to control group.

In eosinophil-guided group, patients will receive prednisone at a dose of 1mg/kg/day for up to 5 days or during the hospital stay if less than 5 days, only if the eosinophil count is> 2%,. Corticosteroid treatment is taken in the morning in patients with NIV, and through the gastric tube in intubated patients.If blood eosinophil count is ≤2%, no corticosteroids are given.

In the control group: A treatment based on prednisone at a daily dose of 1 mg/kg will be routinely administered for a maximum of 5 days, or during the hospital stay, if it is less than 5 days. Corticosteroid treatment is taken in the morning in patients with NIV, and through the gastric tube in intubated patients.

The associated medications will be administered in a standardized way The hypothesis tested is a non-inferiority of the "eosinophil-guided strategy" compared to the standard strategy, with less exposure to corticosteroids.

The primary endpoint is the proportion of unventilated patients at day 6 in study-groups which is set to 50% in the control group. A pre-specified difference <10% would be a non-inferiority margin.

Secondary endpoints are: Number of ICU days alive without ventilatory support within 28 days after recruitment, length of stay in intensive care Unit, the intubation rate in patients initially under NIV, Mortality in the ICU, Hospital mortality.

Safety:New onset of diabetes or worsening of diabetes requiring the start or the increase in insulin therapy, Upper gastrointestinal bleeding (2 g drop of Hb requiring blood transfusion or fibroscopy), Uncontrolled hypertensive crisis requiring the introduction of new antihypertensives, ICU-acquired neuromyopathy, Nosocomial infection, Relapse rate / recurrence defined respectively by the rate of a new hospital consultation and/or admission in the week or the month following index hospitalization.

Sample size calculation: In a non-inferiority study, with an incidence of the event (no ventilation at D6) of 50% in the standard group and this same incidence less than 60% (10% of acceptable difference for non-inferiority) , a power of 80% and alpha error <0.05, it would take 86 patients per arm by anticipating 2% of lost sight (http://www.pharmaschool.co/size8.asp).

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected COPD, and severe acute exacerbation of COPD, corresponding to an acute episode of exacerbation, associated with a hypercapnic respiratory failure (defined by RR> 25 cycles/min, Paco2> 6 kPa, and ph<7.35) requiring ICU admission for ventilatory support.

Exclusion Criteria:

* self-reported or physician-diagnosed asthma,
* life expectancy of less than 30 days,
* allergy to systemic corticosteroids,
* severe mental illness that could not be controlled by medication,
* severe language difficulties or the inability to provide a written informed consent,
* pneumonia or patent infection,
* systemic fungal infections, or
* patients receiving more than 10 mg of chronic systemic corticosteroids (prednisone equivalent) daily.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
proportion of unventilated patients at day 6 | day 6
  patients breathing spontaneously by the 6th day following inclusion

SECONDARY OUTCOMES:
Number of ICU days alive without ventilatory support within 28 days after recruitment | up to 28 days
  number of days without MV by the 28th day
intubation rate in patients initially under NIV | up to 28 days
  NIV failure
hospital death | up to 28 days
  death during hospitalisation

OTHER OUTCOMES:
serious adverse events | up to 28 days
  adverse events of prednisone

CONTACTS AND LOCATIONS:
Locations (4):
- Morocco (2):
  - CHU Arrazi, Marrakesh
  - CHU Ibn Cina, Rabat
- Tunisia (2):
  - CHU Tahar Sfar, Mahdia
  - CHU Fattouma Bourguiba, Monastir

IPD SHARING:
Plan to Share IPD: No